CLINICAL TRIAL: NCT03548246
Title: A Phase 1-2 Multi-Center Study to Assess the Efficacy and Safety of Abiraterone Acetate as Adjunctive Therapy in Pre-Pubescent Children With Classic 21-Hydroxylase Deficiency
Brief Title: Androgen Reduction in Congenital Adrenal Hyperplasia
Acronym: ARCH
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study plan has halted and was withdrawn from the IRB.
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH); University of Michigan (Other); Children's Hospital Los Angeles (Other); Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Perrin C White, MD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 042015-068
Record Dates: First submitted 2015-04-24; First posted 2018-06-07 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Congenital Adrenal Hyperplasia
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital | interventions — Abiraterone Acetate; Hydrocortisone; Fludrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Daily placebo, plus usual maintenance treatment with hydrocortisone and fludrocortisone.
  Interventions: Drug: Placebo; Drug: Hydrocortisone; Drug: Fludrocortisone
- Abiraterone acetate (Experimental): Abiraterone acetate administered daily in dose determined in Phase 1, plus usual maintenance treatment with hydrocortisone and fludrocortisone..
  Interventions: Drug: Abiraterone acetate; Drug: Hydrocortisone; Drug: Fludrocortisone

INTERVENTIONS:
Drug: Abiraterone acetate — Daily oral abiraterone acetate for 2 years. The dose will be specified based on pharmacodynamic data from Phase 1.
  Other Names: Zytiga
  Arms: Abiraterone acetate
Drug: Placebo — Daily placebo for 2 years.
  Arms: Placebo
Drug: Hydrocortisone — Hydrocortisone will be administered at a starting dose of 7-9 mg/M2/d and adjusted as necessary based on 17-hydroxyprogesterone and ACTH levels.
Drug: Fludrocortisone — Fludrocortisone will be administered at the dose the subject was taking a study entry and adjusted as necessary to keep plasma renin in the high normal range.

SUMMARY:
Children with congenital adrenal hyperplasia (CAH) due to 21-hydroxylase deficiency tend to have elevated circulating levels of androgens, which can accelerate skeletal maturation and adversely impact adult height. Additionally, these children require supraphysiologic doses of hydrocortisone to suppress secretion of adrenal androgen precursors, and this treatment can retard linear growth. This study seeks to use oral abiraterone acetate (Zytiga)as an adjunct to approved CAH therapy (oral hydrocortisone and fludrocortisone) for pre-pubescent children with classic 21-hydroxylase deficiency in order to reduce daily requirement of hydrocortisone.

DETAILED DESCRIPTION:
Congenital adrenal hyperplasia (CAH) is an inherited inability to synthesize cortisol in the adrenal gland. More than 90% of cases are cause by deficiency of steroid 21-hydroxylase (CYP21, also termed CYP21A2, P450c21), which is a cytochrome P450 enzyme located in the endoplasmic reticulum. It catalyzes conversion of 17-hydroxyprogesterone (17-OHP) to 11-deoxycortisol, a precursor for cortisol, and progesterone to deoxycorticosterone, a precursor for aldosterone. Aldosterone deficiency may lead to salt wasting with consequent failure to thrive, hypovolemia, shock and if untreated, death in the first few weeks of life. Because patients cannot synthesize cortisol efficiently, the adrenal cortex is stimulated by corticotropin (ACTH) and overproduces cortisol precursors. Some of these precursors are diverted to sex hormone biosynthesis, which may cause signs of androgen excess including ambiguous genitalia in newborn females, rapid postnatal growth in both sexes, and accelerated skeletal maturation and decreased adult height. Patients require supraphysiologic replacement doses of glucocorticoids to suppress the adrenocorticotropic hormone (ACTH)-driven adrenal androgen synthesis. Excessive glucocorticoids are associated with excessive weight gain and slowing of linear growth. It would be desirable in pre-pubertal children to decrease the exposure to excess glucocorticoids while avoiding the adverse effects of inappropriate exposure to androgens. Abiraterone acetate is a prodrug of abiraterone, an irreversible inhibitor of 17α hydroxylase/C17, 20-lyase (cytochrome P450c17 [CYP17]), a key enzyme required for testosterone synthesis. This agent indeed suppresses adrenal androgen secretion in adult women. This Phase 2 will determine if, over 24 months, this treatment retards bone age advancement and thus improves adult height prognosis. The present study is the first clinical trial to explore the utility of abiraterone acetate as a means for decreasing daily requirements for glucocorticoids in pre-pubertal children with 21-hydroxylase deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubescent girls (age 2 years [12 kg] to 8 years inclusive; skeletal age ≤9 years) or boys (age 2 years [12 kg] to 9 years inclusive; skeletal age ≤10 years).
* Confirmed classic 21-hydroxylase deficiency evident by genotype groups A, A1 or B, or by clinical course.
* Requirement for standard of care fludrocortisone (any dose) and ≥10 mg/m2/day of hydrocortisone for at least 1 month prior to the study consent.
* Morning serum androstenedione concentrations >1.5 x ULN after 7 days of dosing with doses of hydrocortisone required for physiologic replacement.
* Informed consent .

Exclusion Criteria:

* Evidence of central puberty: Tanner Stage >2 for breast development in girls or testicular volume >4 mL in boys, or random LH >0.3 mIU/mL.
* Current or history of hepatitis from any etiology.
* Abnormal liver function tests (transaminases>3X ULN).
* Abnormal renal function tests (BUN or creatinine >1.5 ULN).
* Significant anemia (hemoglobin < 12 g/dl).
* Clinically significant ECG abnormality
* A history of a malabsorption syndrome.
* Evidence of active malignancy.
* Co-existent disease that may interfere with linear growth or that requires concomitant therapy that is likely to interfere with study procedures or results.
* Treatment with potentially hepatotoxic medications, CYP2D6, strong inhibitors or inducers of CYP3A4
* Treatment with medications to affect puberty or synthesis of sex steroids, including gonadotropin releasing hormone agonists, aromatase inhibitors, or androgen receptor blockers
* Treatment with growth hormone
* Known allergies, hypersensitivity, or intolerance to abiraterone acetate or its excipients.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Bone age advancement | 104 weeks
  Advancement from baseline in radiographically determined skeletal maturation

SECONDARY OUTCOMES:
Weight | 104 weeks
  Change from baseline, determined every 6 months.
Body mass index Z-score | 104 weeks
  Change from baseline, determined every 6 months.
Predicted adult height | 104 weeks
  Derived from height and radiographically determined skeletal maturation, determined every 6 months
Hydrocortisone dose required to normalize androstenedione levels | 104 weeks
  Hydrocortisone dose (measured as milligrams per meter squared body surface area, per day) will be adjusted in a blinded manner every 3 months by the treating physician to maintain serum androstenedione in the normal range, with increases as necessary to maintain ACTH < 5 times the upper limit of the reference range.
Number of adverse events | 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Perrin C White, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - National Institutes of Health, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Children's Medical Center, Dallas, Texas

REFERENCES:
- [Background] Auchus RJ, Buschur EO, Chang AY, Hammer GD, Ramm C, Madrigal D, Wang G, Gonzalez M, Xu XS, Smit JW, Jiao J, Yu MK. Abiraterone acetate to lower androgens in women with classic 21-hydroxylase deficiency. J Clin Endocrinol Metab. 2014 Aug;99(8):2763-70. doi: 10.1210/jc.2014-1258. Epub 2014 Apr 29. PMID 24780050